CLINICAL TRIAL: NCT04844203
Title: Prevalence of Orthostatic Tremor by Surface Electromyographic Recording in Patients Reporting Unsteadiness
Brief Title: Prevalence of Orthostatic Tremor in Patients With Unsteadiness
Acronym: EMG-SOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191089; 2019-A02976-51 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Orthostatic Tremor; Neuropathy
Keywords: Electroneuromyography; Polygraphy; Unsteadiness; Tremor; Anti-MAG neuropathy; Chronic demyelinating inflammatory neuropathy
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with unsteadiness: Patients with unsteadiness referred for an ENMG
  Interventions: Diagnostic Test: Polygraphy with surface electrodes

INTERVENTIONS:
Diagnostic Test: Polygraphy with surface electrodes — Patients referred for ENMG to the Clinical Physiology Department and complaining of postural unsteadiness will undergo a polygraphy recording using surface electrodes (Natus Medical Incorporated), performed at the end of ENMG

SUMMARY:
Clinical presentation of orthostatic tremor (OT) may be misleading and simply perceived by a postural instability such as in several peripheral neuropathies. In addition, peripheral neuropathies represent the leading cause of pathologies associated with OT. Among patients referred for an electroneuromyogram (ENMG) for peripheral neuropathy and presenting with postural unsteadiness, OT assessment will be systematically performed. Demographic, clinical and polygraphy characteristics of these patients will be analyzed and prevalence of OT in the general population of peripheral neuropathies will be assessed.

DETAILED DESCRIPTION:
Among patients who will be referred for ENMG and exploration of a neuropathy, orthostatic tremor will be investigated systematically.

Main objective and primary endpoint:

* To estimate the prevalence of OT with its 95% confidence interval in the population of patients defined above
* Presence of OT confirmed by surface EMG (polygraphy) in patients with standing instability referred for ENMG.

Secondary objectives and end points

* Determine the demographic, clinical, electrophysiological characteristics of patients with OT; Estimate the prevalence of peripheral neuropathy in patients with OT; Duration of symptoms; Correlation with quantitative neuropathy scores (ISS, MRC, ONLS, R-ODS)
* Age, sex, clinical parameters: symptoms reported by the patient (instability, tremor, weakness, pain, falls), duration, current medications, ISS score, MRC score, ONLS score, R-ODS score) and electrophysiological parameters (mean frequency of OT in Hertz, MUNIX score (number of motor units in the anterior tibialis, calculated by software on the ENMG machine).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* All patients complaining of instability when standing up and referred for an ENMG
* Patient informed and having expressed his non-opposition to participating in the research

Exclusion Criteria:

* Patient's refusal to participate in the study
* Impossibility to stand
* No affiliation to health insurance
* Patients under a legal protection measure or unable to express their will
* Patient under the State Medical Assistance (AME)
* Patient under 18 years old
* Pregnant women, parturients and breast-feeding mothers

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient referred to the Clinical physiology Department for an ENMG (investigation of the neuropathy)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of orthostatic tremor (OT | Day 0
  Prevalence of OT (95% confidence interval) in patients complaining of postural instability and referred for ENMG

SECONDARY OUTCOMES:
Inflammatory Neuropathy Cause and Treatment (INCAT) Sensory Sum Score (ISS) simplified | Day 0
  The ISS ranges from 0 (normal sensation) to 20 (most severe sensory deficit) and is composed of the summation of the following sensation evaluations : pinprick arm grade (range 0-4) ; vibration arm grade (range 0-4) ; pinprick leg grade (range 0-4); vibration leg grade (range 0-4): two-point discrimination grade (range 0-4)
Medical Research Council (MRC) score | Day 0
  The MRC score grades muscle power on a scale of 0 (no detectable contraction) to 5 (normal force, comparable to the healthy side)
Overall Neuropathy Limitations Scale (ONLS) score | Day 0
  The ONLS score is be completed by adding the total of the Arm disability scale score (0-5) and Leg disability scale score (0-7) yielding a total score of 0-12 (higher score indicates higher disability)
Rasch-built Overall Disability Scale (R-ODS) score | Day 0
  R-ODS scale comprising 24 items evaluates the ability to perform daily activities. The answers are rated on a scale of 0 to 48 (with 0 being very poor and 48 being best performance)
OT frequency | Day 0
  OT frequency in Hz
Motor unit number index (MUNIX) | Day 0
  MUNIX is a method for assessment of number of motor units using the compound muscle action potential (CMAP) and surface electromyographic interference pattern (SIP).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie KUBIS, MD, PhD, Principal Investigator — APHP, Lariboisière Hospital
Locations (1):
- APHP Lariboisière Hospital, Clinical Physiology Department, Paris, France